CLINICAL TRIAL: NCT04643197
Title: Effects of Barbed Suture Fascia Closure on Incisional Hernia in Midline Laparotomy for Gynecological Disease (BARBHER)
Brief Title: Effect of Barbed Suture Fascia Closure on Incisional Hernia in Midline Laparotomy for Gynecological Diseases (BARBHER)
Acronym: BARBHER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kidong Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KGOG 4001
Record Dates: First submitted 2020-11-11; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Intervention Model Description: 2*2 factorial design Primary randomization: Barbed suture vs. Non-barbed suture in fascia closure Secondary randomization: subcutaneous drain insertion vs. non-insertion The effect of secondary randomization is one of secondary objectives.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Abdominal fascia will be closed with barbed suture.
  Interventions: Device: Barbed PDS suture (STRATAFIX Symmetric PDS Plus)
- Control (Active Comparator): Abdominal fascia will be closed with non-barbed suture.
  Interventions: Device: Non-barbed PDS suture (PDS Plus)

INTERVENTIONS:
Device: Barbed PDS suture (STRATAFIX Symmetric PDS Plus) — STRATAFIX Symmetric PDS Plus is a barbed suture.
  Arms: Experimental arm
Device: Non-barbed PDS suture (PDS Plus) — Non-barbed suture
  Arms: Control

SUMMARY:
Investigators will compare the incidence of incisional hernia in women who underwent midline laparotomy whose abdominal fascia was closed with barbed suture vs. conventional non-barbed suture.

ELIGIBILITY:
Inclusion Criteria:

* Anticipating midline laparotomy for gynecologic diseases
* ECOG performance status 0 - 2

Exclusion Criteria:

* Previous or current abdominal incisional hernia
* Pregnant
* Previous radiation on abdomen area
* Allergy to PDS or irgacare MP
* Having disease affecting wound healing such as uncontrolled DM, autoimmune vasculitis, liver cirrhosis, coagulopathy
* BMI > 35
* Current or anticipated use of drugs affecting wound healing such as bevacizumab (with 4 week drug free period, bevacizumab user is eligible)
* Abdominal midline laparotomy within 6 months
* Surgery for infection control

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of incisional hernia | from surgery to 1 year
  Incisional hernia till 1 year after surgery

SECONDARY OUTCOMES:
Time-event curve of incisional hernia | from surgery to 1 year
Cumulative incidence of surgical site infection | from surgery to 4weeks
Incidence of wound dehiscence | post-surgery 4weeks
Brief Pain Inventory - Korean (BPI-K) score | Baseline, postoperative day 2, 4
  Pain measured with BPI-K Specifically score (0-10 all domain, higher score mean worse outcome) in domain of worst pain, least pain, average pain, current pain, impact of pain in general activity, mood, work, relationship, ambulation, sleep and happiness
Treatment related adverse event | from surgery to 1 year
NRS | from surgery to postoperative 4 day
  pain captured by NRS in nursing record, 0-10, higher score means more pain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee YJ, Kim NK, Kim K, Choi CH, Lee KH, Lee JM, Lee KB, Suh DH, Kim S, Kim MK, Seong SJ, Lim MC. Effect of fascial closure using barbed sutures on incisional hernias in midline laparotomy for gynecological diseases: A multicenter randomized controlled trial (KGOG 4001). PLoS One. 2025 Nov 19;20(11):e0337036. doi: 10.1371/journal.pone.0337036. eCollection 2025. PMID 41259380
- [Derived] Choi CH, Kim NK, Kim K, Lee YJ, Lee KH, Lee JM, Lee KB, Suh DH, Kim S, Kim MK, Seong SJ, Lim MC. Effects of subcutaneous drain on wound dehiscence and infection in gynecological midline laparotomy: Secondary analysis of a Korean Gynecologic Oncology Group study (KGOG 4001). Eur J Surg Oncol. 2024 Sep;50(9):108484. doi: 10.1016/j.ejso.2024.108484. Epub 2024 Jun 12. PMID 38901293